CLINICAL TRIAL: NCT01201460
Title: Blood Sugar Testing in Dental Patients
Brief Title: DPBRN Blood Sugar Testing in Dental Patients
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other)
Responsible Party: Gregg H. Gilbert, DDS, MBA, Study Chair, The University of Alabama at Birmingham
Other Study IDs: 123961; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus; Hyperglycemia
Keywords: glucose testing
MeSH Terms: conditions — Diabetes Mellitus; Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Glucose testing: Patients participating in this study may be alerted to possible presence of (DM) or pre-(DM) or to inadequate glycemic control. In such a case, they were advised to follow-up with their physician for definitive diagnosis and treatment. Early diagnosis and improved glycemic control may be of significant benefit to the patients' health.

SUMMARY:
The principal goal of this study was to assess the feasibility of plasma glucose testing in private dental practice. A second aim was was to assess prevalence of plasma glucose abnormalities in dental patients seen by (DPBRN) practitioner-investigators.

DETAILED DESCRIPTION:
The specific aims of this study were:

1. To quantify the percentage of (DPBRN) patients who meet the American Diabetes Association screening criteria and to describe the characteristics of these patients.
2. To quantify the acceptability of conducting glucose testing in the dental office and barriers to regular screening, as reported by (DPBRN) patients and practices.

ELIGIBILITY:
Inclusion Criteria:

* adults over the age of 19 who were scheduled for a visit with an exam

Exclusion Criteria:

* patients undergoing continuing treatment where an exam was not part of the visit were not eligible

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The human subjects direclty involved in this study were the patients who had sought dental treatment in the (DPBRN) practitioner-investigators' practices.
Sampling Method: Non-Probability Sample
Enrollment: 498 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Barasch, DMD, MDSc, Principal Investigator — The University of Alabama at Birmingham
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark